CLINICAL TRIAL: NCT01092949
Title: Reference Ranges for Placental Perfusion Using Magnetic Resonance Imaging (MRI)PLACENTIMAGE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P 081111; 2009-A01024-63 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-02-26; First posted 2010-03-25 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Placental Insufficiency
Keywords: Placenta; perfusion; MRI; spin tagging; Gadolinium; placental insufficiency; urinary tract, sexual organs and pregnancy conditions
MeSH Terms: conditions — Placental Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MRI — MRI, 45 minutes
  Other Names: MRI, 45 minutes

SUMMARY:
To evaluate the feasibility of functional MRI method developed in an animal model and to construct normal reference ranges for in vivo placental perfusion using functional MRI. This will be based on imaging studies in patients undergoing termination of pregnancy (TOP) at 16 to 32 weeks' for fetal reason in a tertiary referral center.

DETAILED DESCRIPTION:
Objective:

To evaluate the feasibility of functional MRI method developed in an animal model and to construct normal reference ranges for in vivo placental perfusion using functional MRI. This will be based on imaging studies in patients undergoing termination of pregnancy (TOP) at 16 to 32 weeks' for fetal reason in a tertiary referral center.

Method:

All patients undergoing TOP at 16 to 32 weeks will be offered to participate in this study.

120 patients will be included. 15 per group of weeks of gestation: 16+0-17+6 SA, 18+0-19+6 SA, 20+0-21+6 SA, 22+0-23+6 SA, 24+0-25+6 SA, 26+0-27+6 SA, 28+0-29+6 SA, 30+0-31+6 WG.

MRI will be performed in the same hospital, during hospital stay, within 45 minutes.

Two MRI sequences will be used to measure placental perfusion:

* dynamic sequences using Gd contrast agent.
* " spin tagging ", which do not need any contrast agent. Perfusion will be modelled using compartmental analysis. Reference ranges will be build up by statistical modelling. Gadolinium assays will be performed on amniotic fluid and placental tissue following TOP.

Duration of inclusion: 24 months.

Duration of patient participation: 45 minutes.

Expected results:

* Feasibility in routine practice.
* Reference ranges for placental perfusion.
* Comparison between the two measurements methods.

Adverse outcome measure:

Nausea, vomiting, lack of comfort and other adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years,
* Undergoing TOP for fetal reason,
* Informed signed consent.

Exclusion Criteria:

* Placental adhesion anomaly,
* Growth restriction,
* Contrast agent allergy,
* Absent consent,
* Contraindication of MRI or Gadolinium,
* Renal insufficiency,
* Placental abnormality at pathological examination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing TOP at 16 to 32 weeks will be offered to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Establishment of physiological reference range of placental perfusion | 45 MIN
  Establishment of physiological reference range of placental perfusion

SECONDARY OUTCOMES:
To quantify in vivo and by a not invasive way the microscopic physiological phenomena relative to the placental perfusion and in the local transcapillary exchanges of the placenta | 45 MIN
Comparison between the two measurements methods. | 45 MIN

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Salomon, MCU PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Enfants Malades, Paris, France

REFERENCES:
- [Result] Deloison B, Arthuis C, Benchimol G, Balvay D, Bussieres L, Millischer AE, Grevent D, Butor C, Chalouhi G, Mahallati H, Helenon O, Tavitian B, Clement O, Ville Y, Siauve N, Salomon LJ. Human placental perfusion measured using dynamic contrast enhancement MRI. PLoS One. 2021 Sep 2;16(9):e0256769. doi: 10.1371/journal.pone.0256769. eCollection 2021. PMID 34473740